CLINICAL TRIAL: NCT00551967
Title: Evaluation of the Wear of Vitamin E Treated Polyethylene Components in Primary Total Hip Arthroplasty Using Radiostereometric Analysis (RSA)
Brief Title: Evaluation of the Wear of Vitamin E Treated Polyethylene Components in Primary THA Using RSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Henrik Malchau, Director of Research, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007P000337
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis of Hip; Traumatic Arthritis of Hip
Keywords: clinical outcomes; radiographic outcomes; total hip arthroplasty; survivorship
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E1 polyethylene (Active Comparator): All patients received an E1 polyethylene liner which is the material being monitored in this study.
  Interventions: Procedure: Hip replacement

INTERVENTIONS:
Procedure: Hip replacement — Surgical implantation of hip replacement components for the treatment of osteoarthritis

SUMMARY:
The specific aim of this proposed study is to conduct a prospective RSA clinical study at Massachusetts General Hospital involving 50 patients receiving primary total hip replacements. All patients will receive the vitamin E treated polyethylene acetabular inserts. Short-term femoral head penetration and long-term steady state wear of the polyethylene will be measured using both RSA and Martell analysis techniques. Stability of the acetabular and femoral components will be measured in all patients using RSA analysis. The stability of the cemented femoral stems will be compared to the stability of the cementless femoral components as well as to historic data in the literature. In addition, all patients will complete a self-administered questionnaire to assess the clinical outcome of the surgery and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 20 to 75 years of age
* Subjects requiring primary total hip replacement
* Subjects with diagnosis of osteoarthritis, avascular necrosis, or traumatic arthritis
* Subjects who demonstrate the ability to return to MGH for follow-up for the next five years.

Exclusion Criteria:

* Subjects with limited life span
* Subjects with difficulty in comprehending study protocol for any reason.
* Subjects with inflammatory disease, previous infection or those requiring revision hip surgery.
* Subjects whose bony structures are so small that a femoral head less than 32mm in diameter must be used.
* Subjects whose bony structure deviates substantially from the general norm sufficiently to require non-standard techniques and non-standard implants. Specific examples of these are total dislocation of the hip, severe coxa vera deformity, severe forms of multiple epiphyseal dysplasia
* Subjects with complex disease entities which significantly increase the risks of the surgery such as any major platelet abnormality, hematological disorder, positive for HIV or any other major medical complication which substantially reduces longevity.
* Female subjects that are pregnant or who may suspect they are pregnant or who plan to become pregnant while participating in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Short-term femoral head penetration,long-term steady state wear of polyethylene. Stability of acetabular & femoral components. Clinical questionnaires to assess preop,clinical outcomes,& patient satisfaction. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Malchau, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States